CLINICAL TRIAL: NCT03656250
Title: Assessment of Treatment Response of Nasopharyngeal Cancer Using Simultaneous 18F-FDG-PET and MRI
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-00846
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chemo Patients with Nasopharyngeal cancer: The standard chemoradiation treatment (total 7000 cGy in 35 fractions at 200 cGy/fraction) for 7 weeks with 3 cycles of chemo followed by 3-month chemotherapy.
  Interventions: Diagnostic Test: PET/CT scans

INTERVENTIONS:
Diagnostic Test: PET/CT scans — (approximately 18 mSv/scan) and perform maximum two additional PET/MR scans; one immediately after the first stage of treatment and another one immediately after the second stage if the 3-month chemotherapy is given).

SUMMARY:
The overarching goal of this study is to develop PET/MR techniques for accurate assessment of treatment response during and immediately after chemoradiation therapy. The central hypothesis is that the GMR measured using a simultaneous PET/MR scanner can more accurately detect residual tumor than conventional SUV measures from PET alone. It is important to note that SUV depends on both tumor metabolic rate and tracer delivery, which makes the interpretation of SUV challenging. For instance, inflammatory tissue can have high SUV due to increased vascularity and vascular permeability and cannot be easily differentiated from tumor based on the SUV. Investigators hypothesize that inflammatory tissue will have lower GMR than residual tumor that contain highly proliferating cells with increased expression of glucose transporters (GLUT). Measuring GMR accurately will improve the specificity of PET while maintaining the high sensitivity of PET for detection of residual tumor. In order to test our hypothesis, investigators propose to conduct dynamic PET and MRI scans with NPC patients who are undergoing a conventional two-stage chemoradiation therapy at our institution; the first stage for 7-week chemoradiation therapy followed by the second stage for 3-month chemotherapy. A combination of PET/CT and nasopharynx MRI is currently obtained before the initiation of treatment and 3 months after completion of treatment to assess treatment response.

This study proposes to introduce PET/MR scans at the time of these exams (scan #1 for pre-treatment & scan #4 for 3 months after completion) and to add two additional PET/MR scans in between them; one immediately after the first stage of treatment (scan #2) and another one immediately after the second stage (scan #3). A primary clinical endpoint of this study is the treatment response assessed at 3 months after completion of treatment. A secondary endpoint is 6 month follow-up exam. Complete responder will be determined based on clinical and imaging assessment of residual tumor size at each endpoint.

It is hoped that preliminary data obtained from this study will be useful in planning larger studies to formally investigate the utility of GMR for detection of residual tumor and prediction of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal cancer who are scheduled for chemoradiation therapy at NYU Langone Medical Center or Bellevue hospital are eligible.

Exclusion Criteria:

* Normal MRI exclusion criteria will apply, including those on the following list. A standard MRI safety form will be used to identify potential conditions warranting exclusion.
* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Claustrophobia
* History of seizures
* Diabetes

In addition, patients with GFR < 15 ml/min/1.73m2 or who are on dialysis will be excluded from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (n=20) with nasopharyngeal cancer who are scheduled for chemoradiation therapy are eligible.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolic Rate (GMR) Measured by PET/MR | Day 1
  measured using a simultaneous PET/MR scanner to detect residual tumor
Glucose Metabolic Rate (GMR) Measured by PET/MR | 2 Weeks
  measured using a simultaneous PET/MR scanner to detect residual tumor
Glucose Metabolic Rate (GMR) Measured by PET/MR | 3 Months
  measured using a simultaneous PET/MR scanner to detect residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: Sungheon Kim, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States